CLINICAL TRIAL: NCT01042236
Title: A Phase 2, Randomized, Double-Blind, Multi-Dose, Placebo-Controlled Crossover Study Of The Efficacy Of Fesoterodine In Increasing Urethral Pressure In Stress Urinary Incontinence Patients.
Brief Title: Evaluation Of The Ability Of Fesoterodine To Increase Urethral Pressure In Stress Urinary Incontinence Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: A0221064
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Results first posted 2011-07-01 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Stress Urinary Incontinence
Keywords: Phase 2 stress urinary incontinence Fesoterodine
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — fesoterodine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Fesoterodine

INTERVENTIONS:
Drug: Fesoterodine — Fesoterodine 4 mg and 8 mg and placebo - each dosed for 7 days with 7 day washout between dosing periods
  Other Names: Toviaz

SUMMARY:
The hypothesis under evaluation is that fesotorodine may provide clinical benefit in the treatment of the condition of stress urinary incontinence

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 - 65 years
* SUI symptoms for longer than 3 months
* Subjects must be non-pregnant and not breastfeeding

Exclusion Criteria:

* Disease or medical condition affecting the bladder or urinary tract (other tan stress urinary incontinence)
* Subjects taking medication with effects on the bladder or urinary tract
* Subejcts with medical conditions which could be adversely affected by administration of fesoterodine - gastrointestinal tract disease, glaucoma, hepatic impairment

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Glostrup Hospital, Glostrup Municipality, Denmark

REFERENCES:
- [Derived] Klarskov N, Darekar A, Scholfield D, Whelan L, Lose G. Effect of fesoterodine on urethral closure function in women with stress urinary incontinence assessed by urethral pressure reflectometry. Int Urogynecol J. 2014 Jun;25(6):755-60. doi: 10.1007/s00192-013-2269-6. Epub 2013 Nov 21. PMID 24258099
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221064&StudyName=Evaluation%20Of%20The%20Ability%20Of%20Fesoterodine%20To%20Increase%20Urethral%20Pressure%20In%20Stress%20Urinary%20Incontinence%20Patients

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants randomized to receive sequenced dosing of Fesoterodine 4 milligrams (mg) (A), or Fesoterodine 8 milligrams (B), or Placebo matching study treatment (C). Each dosed for 7 days with a 7 day washout between dosing periods. Dosing sequenced as ABC, ACB, BAC, BCA, CAB, or CBA.
Groups:
- Sequence ABC: Fesoterodine 4 mg (A) tablet administered by mouth (PO) once daily (OD) for 7 days with a 7 day washout period followed by Fesoterodine 8 mg (B) then placebo matching study treatment (C) with 7 day washout between dosing periods.
- Sequence BCA: Fesoterodine 8 mg (B) tablet administered PO OD for 7 days with a 7 day washout period followed by placebo matching study treatment (C) then Fesoterodine 4 mg (A) with 7 day washout between dosing periods.
- Sequence CAB: Placebo matching study treatment (C) tablet administered PO OD for 7 days with a 7 day washout period followed by Fesoterodine 4 mg (A) then Fesoterodine 8 mg (B) with 7 day washout between dosing periods.
- Sequence ACB: Fesoterodine 4 mg (A) tablet administered PO OD for 7 days with a 7 day washout period followed by placebo matching study treatment (C) then Fesoterodine 8 mg (B) with 7 day washout between dosing periods.
- Sequence BAC: Fesoterodine 8 mg (B) tablet administered PO OD for 7 days with a 7 day washout period followed by Fesoterodine 4 mg (A) then placebo matching study treatment (C) with 7 day washout between dosing periods.
- Sequence CBA: Placebo matching study treatment (C) tablet administered PO OD for 7 days with a 7 day washout period followed by Fesoterodine 8 mg (B) then Fesoterodine 4 mg (A) with 7 day washout between dosing periods.
Period: Treatment Period 1
Arm/Group | Sequence ABC | Sequence BCA | Sequence CAB | Sequence ACB | Sequence BAC | Sequence CBA
Started | 3 | 4 | 3 | 5 | 4 | 3
Completed | 3 | 3 | 3 | 5 | 3 | 3
Not Completed | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 1 | 0
Period: Treatment Period 2
Arm/Group | Sequence ABC | Sequence BCA | Sequence CAB | Sequence ACB | Sequence BAC | Sequence CBA
Started | 3 | 3 | 3 | 5 | 3 | 3
Completed | 3 | 3 | 3 | 5 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Sequence ABC | Sequence BCA | Sequence CAB | Sequence ACB | Sequence BAC | Sequence CBA
Started | 3 | 3 | 3 | 5 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive Fesoterodine (4mg) first, Fesoterodine (8mg) first, and Placebo first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 22
Age Continuous [Mean (Standard Deviation); unit: Years] | 47.9 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Opening Urethral Pressure (OUP) at Day 7
Description: OUP measured by urethral reflectometry calculated as the mean of all of the OUP measurements obtained in triplicate at each time point for each participant. Day 7 mean for each treatment period was calculated as the mean of the three measurements taken post-dose on Day 7 of each treatment period separately.
Time Frame: Baseline, Day 7 of each period
Population: Per Protocol Analysis Set (PPAS): all randomized participants who completed the study, received treatment in all 3 study periods until end of treatment visit in the third study period, and had not violated any of the inclusion / exclusion criteria or deviated from the protocol in a way that could affect the outcome of the study.
Measure: Mean (Standard Deviation); unit: centimeter of water (cmH2O)
Groups:
- Fesoterodine (4 mg): Fesoterodine 4 mg tablet administered PO OD for 7 days with a 7 day washout period in either first, second or third treatment period.
- Fesoterodine (8 mg): Fesoterodine 8 mg tablet administered PO OD for 7 days with a 7 day washout period in either first, second or third treatment period.
- Placebo: Placebo matching study treatment for 7 days with a 7 day washout period in either first, second or third treatment period.
Arm/Group | Fesoterodine (4 mg) | Fesoterodine (8 mg) | Placebo
Number analyzed (Participants) | 17 | 17 | 17
centimeter of water (cmH2O)
  Baseline | 49.86 (14.860) | 49.86 (14.860) | 49.86 (14.860)
  Absolute value at Day 7 | 47.92 (12.971) | 49.16 (14.406) | 48.53 (12.859)
  Mean change at Day 7 | -1.94 (4.767) | -0.70 (5.512) | -1.34 (5.178)
Statistical Analysis 1: Comparison: Fesoterodine (8 mg) vs Placebo; Change from baseline (prior to Period 1) at the end of the treatment period was analyzed using an analysis of covariance (ANCOVA) model, with fixed effect terms for sequence, period and treatment, using baseline (prior to Period 1) as a covariate, and participant within sequence as a random effect; Test type: Superiority or Other; p = 0.4907, ANCOVA — A treatment by period interaction term (fixed effect) was included if significant at 10% significance level; Mean Difference (Final Values) = 0.61, 95% CI 2-sided [-1.18 to 2.41], Standard Error of Mean 0.88
Statistical Analysis 2: Comparison: Fesoterodine (4 mg) vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5944, ANCOVA — A treatment by period interaction term (fixed effect) was included if significant at 10% significance level; Median Difference (Final Values) = -0.47, 95% CI 2-sided [-2.27 to 1.32], Standard Error of Mean 0.88

2. Secondary Outcome: Change From Baseline in Closing Urethral Pressure at Day 7
Description: Closing urethral pressure measured by urethral reflectometry calculated as the mean of each of the closing urethral pressure measurements obtained in triplicate at each time point for each participant. Day 7 mean for each treatment period was calculated as the mean of the three measurements taken post-dose on Day 7 of each treatment period separately.
Time Frame: Baseline, Day 7 of each period
Population: PPAS
Measure: Mean (Standard Deviation); unit: cmH20
Arm/Group | Fesoterodine (4 mg) | Fesoterodine (8 mg) | Placebo
Number analyzed (Participants) | 17 | 17 | 17
cmH20
  Baseline | 40.62 (14.379) | 40.62 (14.379) | 40.62 (14.379)
  Absolute value at Day 7 | 37.84 (12.666) | 38.75 (13.172) | 38.66 (11.953)
  Mean change at Day 7 | -2.78 (5.571) | -1.88 (5.475) | -1.96 (5.915)
Statistical Analysis 1: Comparison: Fesoterodine (8 mg) vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9870, ANCOVA — A treatment by period interaction term (fixed effect) was included if significant at 10% significance level; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-1.91 to 1.94], Standard Error of Mean 0.94
Statistical Analysis 2: Comparison: Fesoterodine (4 mg) vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4167, ANCOVA — A treatment by period interaction term (fixed effect) was included if significant at 10% significance level; Mean Difference (Final Values) = -0.78, 95% CI 2-sided [-2.71 to 1.15], Standard Error of Mean 0.94

3. Secondary Outcome: Change From Baseline in Opening Urethral Elastance at Day 7
Description: Opening urethral elastance measured by urethral reflectometry calculated as the mean of each of the opening urethral pressure measurements obtained in triplicate at each time point for each participant. Day 7 mean for each treatment period was calculated as the mean of the three measurements taken post-dose on Day 7 of each treatment period separately.
Time Frame: Baseline, Day 7 of each period
Population: PPAS
Measure: Mean (Standard Deviation); unit: cmH2O/millimeter(mm)^2
Arm/Group | Fesoterodine (4 mg) | Fesoterodine (8 mg) | Placebo
Number analyzed (Participants) | 17 | 17 | 17
cmH2O/millimeter(mm)^2
  Baseline | 1.93 (0.551) | 1.93 (0.551) | 1.93 (0.551)
  Absolue value at Day 7 | 1.66 (0.431) | 1.85 (0.684) | 1.83 (0.690)
  Mean Change at Day 7 | -0.27 (0.396) | -0.08 (0.651) | -0.10 (0.685)
Statistical Analysis 1: Comparison: Fesoterodine (8 mg) vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9403, ANCOVA — A treatment by period interaction term (fixed effect) was included if significant at 10% significance level; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.24 to 0.26], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Fesoterodine (4 mg) vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1881, ANCOVA — A treatment by period interaction term (fixed effect) was included if significant at 10% significance level; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.42 to 0.09], Standard Error of Mean 0.12

4. Secondary Outcome: Change From Baseline in Closing Urethral Elastance at Day 7
Description: Closing urethral elastance measured by urethral reflectometry calculated as the mean of each of the closing urethral pressure measurements obtained in triplicate at each time point for each participant. Day 7 mean for each treatment period was calculated as the mean of the three measurements taken post-dose on Day 7 of each treatment period separately.
Time Frame: Baseline, Day 7 of each period
Population: PPAS
Measure: Mean (Standard Deviation); unit: cmH2O/mm^2
Arm/Group | Fesoterodine (4 mg) | Fesoterodine (8 mg) | Placebo
Number analyzed (Participants) | 17 | 17 | 17
cmH2O/mm^2
  Baseline | 1.85 (0.607) | 1.85 (0.607) | 1.85 (0.607)
  Absolue value at Day 7 | 1.56 (0.347) | 1.74 (0.632) | 1.75 (0.647)
  Mean change at Day 7 | -0.28 (0.391) | -0.10 (0.532) | -0.09 (0.460)
Statistical Analysis 1: Comparison: Fesoterodine (8 mg) vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8602, ANCOVA — A treatment by period interaction term (fixed effect) was included if significant at 10% significance level; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.26 to 0.22], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Fesoterodine (4 mg) vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1271, ANCOVA — A treatment by period interaction term (fixed effect) was included if significant at 10% significance level; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.43 to 0.06], Standard Error of Mean 0.12

5. Secondary Outcome: Incontinence Episode Frequency Per 24 Hours
Description: Incontinence Episode Frequency (IEF) calculated as the average daily total incontinence episodes (stress or urgency) that occurred during the 3 days prior to randomization and the end of each treatment period. Day 7 mean for each treatment period was calculated as the mean daily episode frequency based on the diary completed in the final three days of each treatment period.
Time Frame: Baseline, Day 7 of each period
Population: PPAS
Measure: Mean (Standard Deviation); unit: Episodes per 24 hours.
Arm/Group | Fesoterodine (4 mg) | Fesoterodine (8 mg) | Placebo
Number analyzed (Participants) | 17 | 17 | 17
Episodes per 24 hours.
  Baseline | 1.52 (1.099) | 1.52 (1.099) | 1.52 (1.099)
  Absolute value at Day 7 | 0.71 (0.781) | 0.98 (0.996) | 0.82 (0.698)
  Change at Day 7 | -0.81 (0.866) | -0.54 (1.114) | -0.70 (0.866)

6. Secondary Outcome: Percent Change From Baseline in Incontinence Episode Frequency Per 24 Hours
Description: as for outcome 5
Time Frame: Baseline, Day 7 of each period
Population: PPAS; (n)=only participants with >0 episodes at baseline were to be included in the analysis.
Measure: Median (Full Range); unit: Percent
Arm/Group | Fesoterodine (4 mg) | Fesoterodine (8 mg) | Placebo
Number analyzed (Participants) | 17 | 17 | 17
Percent | -66.67 [-100.0 to 66.7] | -55.56 [-100.0 to 266.7] | -60.00 [-100.0 to 100.0]

7. Secondary Outcome: Stress Incontinence Episode Frequency Per 24 Hours
Description: Stress Incontinence Component of the daily IEF calculated as the average daily number of stress leakage episodes that occurred during the 3 days prior to randomization and the end of each treatment period. Day 7 mean for each treatment period was calculated as the mean daily episode frequency based on the diary completed in the final three days of each treatment period.
Time Frame: Baseline, Day 7 of each period
Population: PPAS
Measure: Mean (Standard Deviation); unit: Episodes per 24 hours.
Arm/Group | Fesoterodine (4 mg) | Fesoterodine (8 mg) | Placebo
Number analyzed (Participants) | 17 | 17 | 17
Episodes per 24 hours.
  Baseline | 1.44 (1.052) | 1.44 (1.052) | 1.44 (1.052)
  Absolute value at Day 7 | 0.69 (0.759) | 0.98 (0.996) | 0.82 (0.698)
  Change at Day 7 | -0.75 (0.812) | -0.46 (1.043) | -0.62 (0.897)

8. Secondary Outcome: Percent Change From Baseline in Stress Incontinence Episode Frequency Per 24 Hours
Description: as for outcome 7
Time Frame: Baseline, Day 7 of each period
Population: PPAS; (n)=only participants with >0 episodes at baseline were to be included in the analysis.
Measure: Median (Full Range); unit: Percent
Arm/Group | Fesoterodine (4 mg) | Fesoterodine (8 mg) | Placebo
Number analyzed (Participants) | 17 | 17 | 17
Percent | -66.67 [-100.0 to 100.0] | -55.56 [-100.0 to 266.7] | -60.00 [-100.0 to 200.0]

9. Secondary Outcome: Urgency Urinary Incontinence Episode Frequency Per 24 Hours
Description: Urgency Urinary Incontinence Component of the daily IEF calculated as the average daily number of urgency leakage episodes that occurred during the 3 days prior to randomization and the end of each treatment period. Day 7 mean for each treatment period was calculated as the mean daily episode frequency based on the diary completed in the final three days of each treatment period.
Time Frame: Baseline, Day 7 of each period
Population: PPAS
Measure: Mean (Standard Deviation); unit: Episodes per 24 hours.
Arm/Group | Fesoterodine (4 mg) | Fesoterodine (8 mg) | Placebo
Number analyzed (Participants) | 17 | 17 | 17
Episodes per 24 hours.
  Baseline | 0.08 (0.251) | 0.08 (0.251) | 0.08 (0.251)
  Absolute value at Day 7 | 0.02 (0.081) | 0.00 (0.000) | 0.00 (0.000)
  Change at Day 7 | -0.06 (0.243) | -0.08 (0.251) | -0.08 (0.251)

10. Secondary Outcome: Percent Change From Baseline in Urgency Urinary Incontinence Episode Frequency Per 24 Hours
Description: as for outcome 9
Time Frame: Baseline, Day 7 of each period
Population: PPAS; (n)=only subjects with >0 participants at baseline were to be included in the analysis.
Measure: Median (Full Range); unit: Percent
Arm/Group | Fesoterodine (4 mg) | Fesoterodine (8 mg) | Placebo
Number analyzed (Participants) | 2 | 2 | 2
Percent | -50.00 [-100.0 to 0.0] | -100.00 [-100.0 to -100.0] | -100.00 [-100.0 to -100.0]

11. Secondary Outcome: Plasma 5-hydroxymethyl Tolterodine (5- HMT) Concentration
Description: Plasma 5-HMT concentration data pre and post reflectometry following multiple doses of fesoterodine 4 mg OD and fesoterodine 8 mg OD. Day 7 mean for each treatment period was calculated as the mean of the three measurements taken post-dose on Day 7 of each treatment period separately. Summary statistics were to be calculated by setting concentration values below the lower limit of quantification (LLQ = 0.02 ng/mL) to zero. Summary statistics were not to be presented if number of observations above lower limit of quantification (NALQ) = 0.
Time Frame: Baseline, Day 7 of each period
Population: Full Analysis Set (FAS): all randomized subjects who had taken at least one dose of study treatment; (n)=number of participants with observations (non-missing concentrations)
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Fesoterodine (4 mg) | Fesoterodine (8 mg)
Number analyzed (Participants) | 18 | 18
nanogram/milliliter (ng/mL)
  Pre-Reflectometry (n=18, 18) | 2.303 (1.2798) | 4.902 (2.1554)
  Post-Reflectometry (n=18, 17) | 2.185 (1.1970) | 4.971 (1.8195)

ADVERSE EVENTS:
Time Frame: Baseline (Period 1 / Day 1) up 28 days after last dose of study treatment
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Fesoterodine (4 mg) | Fesoterodine (8 mg) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/22 | 0/20
Other Adverse Events (participants affected / at risk) | 8/20 | 17/22 | 8/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fesoterodine (4 mg) (N=20) | Fesoterodine (8 mg) (N=22) | Placebo (N=20)
Hypotension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fesoterodine (4 mg) (N=20) | Fesoterodine (8 mg) (N=22) | Placebo (N=20)
Dry Eye (Eye disorders) | 0 | 1 | 0
Vitreous disorder (Eye disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 3 | 12 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 4 | 5 | 2
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Dysmenorrhea (Reproductive system and breast disorders) | 1 | 1 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.